CLINICAL TRIAL: NCT01805258
Title: Efficacy and Safety of Concomitant Use of Nevirapine and Rifampicin in Antiretroviral Naive Patients Co-infected With HIV and Tuberculosis in India.
Brief Title: Efficacy and Safety of Concomitant Use of Nevirapine and Rifampicin With HIV-TB
Acronym: "NVP"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: National AIDS Control Organisation (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKS/NACO-1/2006-07
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: HIV/TB Co-infection
Keywords: India; Nevirapine; Rifampicin; Efavirenz; HIV; TB
MeSH Terms: interventions — Nevirapine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention 2: Nevirapine (Experimental): HIV and Tuberculosis co-infected patients on standard dose nevirapine (Intervention) based ART and Rifampicin based ATT.
  Interventions: Drug: Nevirapine
- Intervention 2: Efavirenz (Active Comparator): HIV and Tuberculosis co-infected patients on standard dose Efavirenz(Intervention)based ART and Rifampicin based ATT.
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Nevirapine — The regimen containing Nevirapine: 3TC/ZDV 150/300 mg 1 tablet BID + NEVIRAPINE 200 mg qD for 2 weeks then 200mg BID
  Other Names: NEV-Nevirapine
  Arms: Intervention 2: Nevirapine
Drug: Efavirenz — The regimen containing Efavirenz: 3TC/ZDV 150/300 mg 1 tablet BID + EFAVIRENZ 600 mg qD
  Other Names: EFV: Efavirenz
  Arms: Intervention 2: Efavirenz

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Nevarapine and Rifampicin vs Efavirenz and Rifampicin in antiretroviral naive patients co-infected with HIV and TB and to investigate whether Rifampicin co-administration in clinical practice leads to a clinically relevant decrease of Nevirapine plasma concentrations in Indian patients co-infected with HIV and Tuberculosis and to characterize drug-associated toxicities (especially hepatic).

DETAILED DESCRIPTION:
Drug interactions complicate concurrent treatment of HIV and Mycobacterium tuberculosis co-infection. Drug therapy for HIV and tuberculosis each consists of combined regimens with three or four drugs. Tuberculosis (TB) is the most significant co-infection of HIV patients in resource-limited settings. Application of antiretroviral (ARV) therapy in co-infected patients will require care providers who are appropriately trained in the use of ARV and TB drugs. Over 40 million people worldwide are currently living with HIV/AIDS, of which 90% live in the developing world, co-infected with TB. There are an estimated 12 million persons with TB/HIV co-infection. According to UNAIDS estimates, 5 million people have acquired HIV/AIDS in 2003. India is estimated to have 5.1 million HIV individuals by the end of 2002. TB is among the most frequent HIV-related opportunistic infections in developing countries, and is associated with substantial morbidity and mortality. In India, there were estimated 1.85 million HIV individuals co-infected with HIV and TB. In patients infected with both HIV and TB, the lifetime risk of developing the active tuberculosis has been estimated to be at least 60%, compared to approximately 10% in persons infected with TB who do not have HIV infection. It is well established that HIV increases the risk for TB (acquisition, reactivation and reinfection), alters its clinical presentation, and reduces survival compared to patients with TB and no HIV infection. Multiple epidemiologic studies have shown that co-infection with TB results in reduced survival, increased risk for opportunistic infections and elevations in HIV replication. Increased HIV replication is attributed to activation of latently infected cells and promotion of infection in uninfected lymphocytes and macrophages. HIV genetic diversity is also increased in the presence of active TB infection. Mortality rates in HIV-infected patients with TB are extraordinarily high in resource- limited settings. Therefore, it is essential to treat patients with HIV and TB co-infection for both infections. In India large numbers of HIV positive patients suffering with HIV/Tuberculosis co-infection. However, limited data are available for concomitant use of Nevirapine and Rifampicin in patients co-infected with HIV and Tuberculosis in India. No concrete data available about whether or not Nevirapine and Rifampicin can be safely co-administered without the plasma concentration of Nevirapine falling below therapeutic levels.

Rifamycins are frequently used for the treatment of tuberculosis. Rifamycins can interact with several antiretrovirals. In decreasing order of potency, rifampin, rifapentine and rifabutin have an inducing effect on drug metabolism mediated through cytochrome P450 isoenzyme 3A4 (CYP3A4). Non-nucleoside reverse transcriptase inhibitors and protease inhibitors are metabolized through CYP3A4 and thus the plasma concentrations of these antiretrovirals may decrease in the presence of rifamycins. Additionally, the non-nucleoside reverse transcriptase inhibitors are metabolized by CYP2B6. Drug-drug interactions may lead to suboptimal drug exposure, loss of viral suppression and selection of resistant HIV strains. Interactions between nucleoside analogue reverse transcriptase inhibitors and rifamycins occur at the level of glucuronidation and amination, as was described between rifampin or rifabutin and zidovudine, but is not considered to be clinically significant.

Coinfection of HIV-1 and tuberculosis mainly concerns developing countries like India where both infections are epidemic. Access to antiretrovirals may be difficult in developing countries because of limited availability or high cost. To improve pricing and accessibility, generic antiretroviral agents are manufactured in countries such as Brazil, India, Thailand and South Africa. Fixed-dose combinations of these generic agents are widely used as well. The most often-used generic fixed-dose combination is a twice-daily regimen with stavudine, lamivudine and nevirapine. Fixed-dose combinations are attractive regimens for patient care. Adherence to therapy may be improved because of low pill burden and the reduced possibility of incorrect dosing. Furthermore, the fixed-dose combinations simplify drug logistics. Compact drug quantities facilitate storage and distribution to hospitals, pharmacies and patients. Important for resource constraint settings is that fixed-dose combinations make improvements in public health care management possible. With respect to treatment of HIV/tuberculosis-coinfected patients, a clinically significant drug-drug interaction may be expected when nevirapine and rifamycin are co-administered. Treatment with rifabutin is preferred because of a more favourable interaction profile, but in most developing countries rifabutin is not available or too expensive. Tuberculosis treatment with a regimen that includes rifampicin is usually the only option. Reports in the literature have shown decreases in nevirapine plasma concentrations ranging from 31% to 58%. Rifampicin plasma concentrations are not influenced by nevirapine. Low nevirapine plasma concentrations may negatively affect virological outcome of antiretroviral therapy. Previous studies have documented higher plasma concentrations of nevirapine in Thai patients compared with patients in other countries, suggesting that even though the concomitant use of rifampicin lowers the nevirapine levels considerable, still most patients would still retain nevirapine plasma concentrations above a concentration of 3.1mg/l. The present study will be performed to investigate whether rifampicin co-administration in clinical practice leads to a clinically relevant decrease of nevirapine plasma concentrations in North Indian patients co-infected with HIV/Tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection, documented by ELISA test
2. Adult patients
3. Patients co-infected with HIV and Tuberculosis
4. Concomitant use of Nevirapine and Rifampicin in patients co-infected with HIV and Tuberculosis
5. ART Naïve patients

Exclusion Criteria:

1. Allergy/hypersensitivity to any study drug(s).
2. Prior history of documented drug-resistant TB.
3. Pregnancy
4. Patients with alanine aminotransferase or aspartate aminotransferase levels more than five times the upper limit of normal.
5. Chronic liver disease due to cirrhosis of liver, hepatitis B & C virus infection.
6. Chronic alcoholic.
7. Non-complaint patients.
8. Migrant patients.
9. Serious form of pulmonary or extrapulmonary tuberculosis e.g. severe haemoptysis and unconscious patients
10. Concomitant diabetes mellitus.
11. Epilepsy
12. Patients on other immunosuppressive therapy.
13. Malignancy other than Kaposi's Sarcoma requiring therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Virological suppression at 48 weeks. | 5 years
  All patients underwent a detailed physical examination. Their body weight and height will be measured and their body mass index (BMI) was calculated. Haemoglobin, complete blood counts, erythrocyte sedimentation rate, fasting blood glucose, renal function tests, liver function tests, serum albumin, serum uric acid and routine urinalysis will be done for all patients.
  Patients will be assessed at day 14 after the start of ART, then at day 28, 42 and every 4 weeks thereafter through 48 weeks. A complete haemogram, liver and kidney function tests will be obtained at all these visits. CD4 counts will be measured at 8 weeks, 24 weeks and 48 weeks after the start of ART. HIV plasma viral load will be measured at baseline, at 24 weeks and at the end of 48 weeks only in the cases. Trough nevirapine concentrations were assessed at day 14, day 28, day 42 and day 180, 12 hours after the evening dose of nevirapine.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events especially Hepatotoxicity as a measure of Safety. | 5 years
  Drug associated toxicities specially hepatitis were assessed in the subjects by performing liver function tests every 4 weeks during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD, Ph.D, Principal Investigator — All India Institute of Medical Science, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, India

REFERENCES:
- [Derived] Sinha S, Gupta K, Tripathy S, Dhooria S, Ranjan S, Pandey RM. Nevirapine- versus Efavirenz-based antiretroviral therapy regimens in antiretroviral-naive patients with HIV and Tuberculosis infections in India: a multi-centre study. BMC Infect Dis. 2017 Dec 11;17(1):761. doi: 10.1186/s12879-017-2864-0. PMID 29228918
- [Derived] Sinha S, Raghunandan P, Chandrashekhar R, Sharma SK, Kumar S, Dhooria S, Ekka M, Velpandian T, Ranjan S, Ahmad H, Samantaray JC, Venkatesh S, Rewari BB, Khan NH, Pandey RM. Nevirapine versus efavirenz-based antiretroviral therapy regimens in antiretroviral-naive patients with HIV and tuberculosis infections in India: a pilot study. BMC Infect Dis. 2013 Oct 17;13:482. doi: 10.1186/1471-2334-13-482. PMID 24134449